CLINICAL TRIAL: NCT07294534
Title: An Open-Label, Randomized, Multicenter Phase II/III Clinical Study to Evaluate the Efficacy and Safety of HLX87 (HER2 ADC) in Combination With HLX22 (Recombinant Humanized Anti-HER2 Monoclonal Antibody Injection) or Pertuzumab vs. TCbHP in the Neoadjuvant Therapy of HER2-Positive Early or Locally Advanced Breast Cancer
Brief Title: A Phase II/III Clinical Study to Evaluate the Efficacy and Safety of HLX87in Combination With HLX22 or Pertuzumab in the Neoadjuvant Therapy of HER2-Positive Bresat Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX87-BC002
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: HER2 + Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HLX87+ HLX22 (Experimental): Patients will receive the treatment once every 3 weeks (Q3W), for 8 cycles.
  Interventions: Drug: HLX87+HX22
- HLX87+ Pertuzumab (Experimental): Patients will receive the treatment once every 3 weeks (Q3W), for 8 cycles.
  Interventions: Drug: HLX87 + Pertuzumab
- TCbHP (Active Comparator): Patients will receive the treatment once every 3 weeks (Q3W), for 6cycles.
  Interventions: Drug: TCbHP

INTERVENTIONS:
Drug: HLX87+HX22 — HLX87 is a novel HER2-targeted ADC with a similar mechanism of action to trastuzumab deruxtecan. HLX22 is a novel monoclonal antibody targeting HER2
  Arms: HLX87+ HLX22
Drug: HLX87 + Pertuzumab — HLX87 is a novel HER2-targeted ADC with a similar mechanism of action to trastuzumab deruxtecan.
  Arms: HLX87+ Pertuzumab
Drug: TCbHP — Docetaxel +Carboplatin+Trastuzumab+Pertuzumab+
  Arms: TCbHP

SUMMARY:
The study is being conducted to evaluate the clinical efficacy of HLX87 in combination with HLX22 or pertuzumab vs. TCbHP in the neoadjuvant therapy of HER2-positive early or locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have a full understanding of the study content, process, and possible adverse reactions before the study, and sign the informed consent form (ICF); voluntarily participate in the study; be able to complete the study as per protocol requirements; 2. Aged ≥ 18 years at the time of signing the ICF, male or female; 3. Primary breast cancer meeting the following criteria:

  1. Histologically confirmed invasive breast cancer;
  2. Clinical stage (assessed by mammography or MRI): T0-4 (including inflammatory breast cancer), N1-3, M0; or ≥ T3, N0, M0 (according to AJCC 8th edition);
  3. HER2-positive as determined by the central laboratory, defined as IHC 3+ or IHC 2+ and ISH-positive;
  4. For unifocal and multifocal tumors (i.e., more than one tumor, all confined to the same quadrant as the primary tumor), at least 1 lesion should be sampled and confirmed as HER2-positive by the central laboratory;
  5. For multi-centric tumors (i.e., multiple tumors involving two or more quadrants of the breast), 1 lesion should be sampled from each affected quadrant and confirmed as HER2-positive by the central laboratory, and all tested quadrants must be confirmed as HER2-positive;
  6. Positive or negative for hormone receptors HR (including estrogen receptor [ER] and progesterone receptor [PgR]) as determined by the central laboratory.

Note: According to ASCO-CAP guidelines, HR-positive is defined as: ER and/or PgR ≥ 1% cells have nuclear staining; HR-negative is defined as: ER < 1% cells have nuclear staining and PR < 1% cells have nuclear staining.

During the screening period, unstained tumor sections should be provided to the central laboratory for relevant tests according to the laboratory manual.

4. Consent for surgery after neoadjuvant therapy. 5. Baseline left ventricular ejection fraction (LVEF) ≥ 55% measured by echocardiography (ECHO) or multi-gated acquisition (MUGA) scan (within 28 days prior to the first dose).

6. No prior systemic anti-tumor treatment for this current breast cancer (including systemic chemotherapy, molecular targeted drug therapy, biological therapy, and other investigational medicinal products).

7. ECOG PS score of 0-1 within 7 days prior to the first dose. 8. Hepatitis B surface antigen (HBsAg) (-) and hepatitis B core antibody (HBcAb) (-). In case of HBsAg (+) or HBcAb (+), hepatitis B virus deoxyribonucleic acid (HBV-DNA) must be < 2500 copies/mL or 500 IU/mL or within the reference range of the site.

9. HCV antibody (-); subjects with HCV antibody (+) must have a negative HCV-RNA test result to be enrolled. Subjects with HBV/HCV co-infection shall be excluded (positive for HBsAg or HBcAb and positive for HCV antibody) 10. HIV antibody (-). 11. Have adequate organ function as defined by the following criteria (no blood transfusions, or treatment with albumin, recombinant human thrombopoietin or colony-stimulating factor [CSF] within 14 days prior to the first dose in this study) 12. Female subjects of childbearing potential must have a negative serum pregnancy test result within 7 days prior to the first dose. Female subjects of childbearing potential and male subjects with female partners of childbearing potential are required to take a medically approved contraceptive measure (e.g., intra-uterine contraceptive device, contraceptive pills, or condoms) during the study treatment period and for at least 7 months after the last dose of study treatment.

Exclusion Criteria:

* 1. Past medical history of invasive breast carcinoma. 2. Stage IV (metastatic) breast cancer (per AJCC 8th edition). 3. History of any second malignancy within 3 years prior to signing the ICF, except for early-stage malignancies (carcinoma in situ or stage I tumors) that have received radical treatment, such as non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, ductal carcinoma in situ of the breast, and papillary thyroid carcinoma.

  4. With serious heart disease or medical history, including but not limited to the following conditions:
  1. Any previous and current heart failure or systolic dysfunction meeting the NYHA criteria;
  2. High-risk uncontrollable arrhythmia: atrial tachycardia with resting heart rate > 100 beats/min, significant ventricular arrhythmia (such as ventricular tachycardia), or high-grade atrioventricular block (such as Mobitz II second-degree atrioventricular block or third-degree atrioventricular block);
  3. Unstable angina or angina requiring antianginal medication
  4. History of transmural myocardial infarction shown by ECG
  5. Clinically significant cardiac valvular disease;
  6. Poorly controlled hypertension (with systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg).

  5. Cerebrovascular accident within 6 months prior to the first dose. 6. Use of immunosuppressants within 14 days prior to the first dose, except for intranasal and inhaled corticosteroids, systemic corticosteroids with a dose of less than 10 mg/day of prednisone/prednisolone or equivalent.

  7. Active systemic infection requiring intravenous antibiotics, antivirals, or antifungals within 7 days prior to the first dose.

  8. History of (non-infectious) pneumonitis/interstitial lung disease (ILD) that required steroids, current presence of pneumonitis/ILD, or suspected pneumonitis/ILD cannot be ruled out by imaging during the screening period.

  9. Have a lung-specific intercurrent clinically significant illness including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary embolism within 3 months prior to dosing, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive pulmonary disease, significant pleural effusion etc.), any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis etc.), and/or prior pulmonary resection.

  10. Presence of active tuberculosis. 11. Have received treatment with live attenuated vaccines within 30 days prior to the first dose. Note: If the patient is enrolled, live vaccines should not be administered during the study and within 30 days after the last study treatment.

  12. Participation in other clinical studies within 30 days prior to signing the informed consent form. Unless the clinical study is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

  13. Known history of severe anaphylaxis to macromolecular protein preparations, hypersensitivity to any component in the formulation of the investigational product, or severe hypersensitivity to any excipients of investigational product.

  14. Have received major surgery within 28 days prior to the first dose. In this study, a major surgery is defined as any surgery which requires at least 3 weeks of postoperative recovery time before receiving the study treatment. Local radiotherapy, radiofrequency ablation, and interventional therapy (excluding previous diagnostic biopsy) within 2 weeks prior to the first dose.

  15. Known history of abuse of psychotropic drugs or drug addiction. 16. Pregnant or lactating women. 17. Other factors, as determined by the investigator, which may result in premature discontinuation of treatment. For example, other serious medical conditions (including mental illnesses) requiring concomitant treatment, serious laboratory abnormalities, family or social factors, and other conditions that may affect the safety of the subjects or the collection of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 817 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
• Total pathologic complete response (tpCR) rate | up to 24 weeks
  as assessed by the Independent Review Committee (IRC). tpCR is defined as the absence of histological evidence of malignancy in both the primary lesion of breast cancer and regional lymph nodes (i.e., ypT0/Tis, ypN0 in the AJCC staging system, 8th edition).

SECONDARY OUTCOMES:
• tpCR rate assessed by the study site | up to 24 weeks
• Breast pathologic complete response (bpCR) rate | up to 24 weeks
Objective response rate (ORR) | up to 24 weeks
Incidence and severity of adverse events (AEs) | time from the date of the first dose of study drug until the date of death from any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Shao, Dr, Principal Investigator — Fudan University